CLINICAL TRIAL: NCT03658720
Title: Randomised, Open Label, Single Dose, 2-way Crossover Study to Evaluate Oral Disintegration Time of a Single Nurofen Ibuprofen Orodispersible Tablet (ODT) and Two Nurofen Ibuprofen ODTs (200mg Ibuprofen Acid), in Fasted Healthy Volunteers
Brief Title: Nurofen Ibuprofen Orodispersible Tablet Disintegration Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was not feasible as designed to allow for appropriate completion
Sponsor: Reckitt Benckiser Healthcare (UK) Limited (Industry)
Collaborators: Simbec Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 0414106
Record Dates: First submitted 2018-04-26; First posted 2018-09-05 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-04

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single tablet (Experimental): Ibuprofen acid ODT: 1x200mg dose. Administered without water after the subject has swallowed (with oral cavity rinsing) 20 mL of water. This was following a fasting period of 2 hours 15 minutes (± 15 minutes). The fasting period started after the subject consumed a standardised light meal/snack.
  Interventions: Drug: 200 mg Ibuprofen acid orodispersible tablet
- Two tablets (Experimental): Ibuprofen acid ODTs: 2x200mg dose. Administered without water after the subject has swallowed (with oral cavity rinsing) 20 mL of water. This was following a fasting period of 2 hours 15 minutes (± 15 minutes). The fasting period started after the subject consumed a standardised light meal/snack.
  Interventions: Drug: 200 mg Ibuprofen acid orodispersible tablet

INTERVENTIONS:
Drug: 200 mg Ibuprofen acid orodispersible tablet — orodispersible tablet
  Other Names: Meltlet; Nurofen

SUMMARY:
Disintegration time is an important quality attribute of ODTs, and the evaluation of disintegration time is positioned as a key step in formulation development, manufacturing, and clinical practice. The standard recommended over-the counter dose of 200mg Nurofen ibuprofen ODT is one (200mg) to two (400mg) tablets. To reflect this, the disintegration time of both one (200mg) and two (400mg) tablets will be assessed in this study.

Studies have been performed assessing in vivo ODT disintegration time and have created standardised oral conditions by giving water prior to dosing, to moisten/wet the mouth. In this study it is therefore necessary to standardise the oral conditions as much as possible, despite the interpersonal variability, to measure the time it takes for the ODT to disintegrate. For this study, 20 mL of water is swallowed prior to dosing to standardise oral conditions. Thirty-three healthy volunteers are required to be randomised into the study, to allow evaluable data to be obtained for 30 subjects. Subjects are given a light meal/snack and then fast for 2 hours 15 minutes (± 15 minutes) before dosing, in order to bring the oral cavity environment as close as possible to standard levels and to minimise variability in salivation. Directly before dosing, subjects drink (with oral cavity rinsing) 20 mL of water. Subjects are dosed according to the sequence they have been randomised and the ODT disintegration time assessed.

Following the first dose, subjects complete a washout period of a minimum of 4 hours, in accordance with the recommended posology, before receiving the second dose. During this washout period, subjects are given a second light meal/snack (the same as the previous light meal/snack), timed to allow subjects to fast for 2 hours 15 minutes (± 15 minutes) before the second dose. Directly before the second dose, subjects drink (with oral cavity rinsing) 20 mL of water. Subjects then receive the alternative dose to the dose they received during the first assessment, in accordance with the randomisation sequence.

Following completion of the disintegration assessments, or upon subject withdrawal, subjects are asked whether they are experiencing any symptoms or complaints. Any AEs are recorded in the CRF and followed up as necessary by the Investigator. Subjects then leave the clinic.Subjects are contacted by the Investigator (or designee) from 24 to up to 48 hours to ensure any AEs are captured.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects who have given written informed consent.
2. Age: ≥ 18 years ≤ 50 years.
3. Body Mass Index (BMI) of ≥ 18.5 and ≤ 30 kg/m2.
4. Healthy as determined by past medical history, physical examination and vital signs at screening.

Exclusion Criteria:

1. A history of allergy or intolerance (including angioedema, urticaria, bronchospasm, reflux symptoms and rhinitis) related to treatment with ibuprofen, aspirin or other NSAIDs, or the excipients of the formulations.
2. A history (treated or untreated) of an oral condition affecting salivation and mouth dryness (e.g. dry mouth, hypersalivation)
3. A history of hepatic or renal impairment, hepatic dysfunction, cardiovascular disease, cerebrovascular problems or high blood pressure.
4. A history of asthma.
5. A history of peptic or duodenal ulcers or upper gastro-intestinal bleed, or other significant gastro-intestinal disorders (including gastro-oesophageal reflux symptoms or gastritis) ulceration, perforation or haemorrhage.
6. A history of coagulation disorder or susceptibility to bleeding
7. A current or recent (within 2 months) oral issue, which in the opinion of the Principal Investigator could interfere with the study (e.g. mouth ulcers, aphthous ulcers, herpetic disease, oral candidiasis, burning mouth syndrome, geographic tongue, oral swellings, sores or lesions.
8. Those currently suffering from dehydration
9. A current or history of oral piercing.
10. A current or recent history (within one year of the study) of alcohol abuse or significant abuse/misuse of any legal or illegal drugs, substances and solvents
11. Those with a positive screen/test for drugs of abuse and/or alcohol
12. Those who consume more than 14 units of alcohol per week, and where this consumption is spread over less than 3 days, or those who regularly (weekly) consumed excessive amounts of alcohol (>8 units for men and >6 units for women in one consumption, excessive amounts as defined by the UK National Office of Statistics)
13. Those who had consumed alcohol within the 24 hours before enrolment onto the study.
14. Those who had regularly consumed excessive quantities of caffeine (>6 cups of tea, coffee or cola per day), according to the Investigator's judgment.
15. Those who had consumed caffeine-containing food and drinks within the 24 hours before enrolment onto the study.
16. Those who had performed strenuous exercise within the 24 hours before enrolment onto the study.
17. Those who currently or have recently (within last 6 months) use/d tobacco or nicotine containing products.
18. Those who have used any herbal/vitamin or fish oil supplement in the 7 days prior to enrolment
19. Those who have used any OTC or prescription medications (except hormonal contraceptives) in the 7 days prior to enrolment
20. Those who have used ibuprofen with concomitant aspirin or other NSAIDs including cyclooxygenase-2 selective inhibitors and any drugs that should be used with caution, in combination with ibuprofen as per the SmPC, in the 7 days prior to enrolment (or longer if stated within the SmPC)
21. Those previously randomised into this study.
22. Those who are an employee at the study site.
23. Those who are a partner or first-degree relative of the Investigator or other employees.
24. Those who have participated in any taste testing study within 3 days of the screening visit.
25. Those who have participated in a clinical trial involving consumption of an investigational medicinal product within 3 months of dosing or a study with a marketed compound in the last month before dosing.
26. Those unable in the opinion of the Investigator to comply fully with the study requirements.
27. Women who are pregnant or breast feeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2017-12-21 (Actual)

PRIMARY OUTCOMES:
Tablet disintegration time | Time of dosing to complete disintegration of the tablet being achieved (2 doses; single assessment day)
  Time to complete tablet disintegration in seconds

SECONDARY OUTCOMES:
Number of Adverse Events | Up to follow up (24-48 hours after assessment day)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Research Director, Clinical Research, Study Director — Reckitt Benckiser Healthcare (UK) Limited
Locations (1):
- Simbec Reseach Limited, Merthyr Tydfil, United Kingdom

IPD SHARING:
Plan to Share IPD: No